CLINICAL TRIAL: NCT00270894
Title: Pilot Trial of Sequential Dose-Dense Neoadjuvant Chemotherapy Plus Herceptin in HER2 Positive Stage II-III Breast Cancer Patients
Brief Title: Neoadjuvant Chemotherapy + Herceptin in HER2 Positive Stage II-III Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACORN ALSSNBC0401
Record Dates: First submitted 2005-12-28; First posted 2005-12-29 (Estimated); Results first posted 2012-03-12 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Breast Neoplasm
Keywords: neoadjuvant chemotherapy; HER2 positive breast cancer; stage II - III breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Docetaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant therapy (Experimental): Neoadjuvant therapy will consist of epirubicin (100 mg/m^2) + cyclophosphamide (600 mg/m^2) every 2 weeks for 4 cycles; followed by a 3-week break; followed by docetaxel (75 mg/m^2) every 2 weeks for 4 cycles + trastuzumab (6 mg/kg [loading dose] once then 4 mg/kg [maintenance dose]) every 2 weeks for 4 treatments.
  Interventions: Drug: epirubicin; Drug: cyclophosphamide; Drug: docetaxel; Drug: trastuzumab

INTERVENTIONS:
Drug: epirubicin — epirubicin (100 mg/m^2) every 2 weeks for 4 cycles
  Other Names: Ellence®
Drug: cyclophosphamide — cyclophosphamide (600 mg/m^2) every 2 weeks for 4 cycles
  Other Names: Cytoxan
Drug: docetaxel — docetaxel (75 mg/m^2) every 2 weeks for 4 cycles
  Other Names: Taxotere®
Drug: trastuzumab — trastuzumab (6 mg/kg [loading dose] once then 4 mg/kg [maintenance dose]) every 2 weeks for 4 treatments
  Other Names: Herceptin®

SUMMARY:
The purpose of this study is to evaluate the effectiveness and tolerability of the combination of the following medications given every two weeks in HER2 positive breast cancer patients:

* trastuzumab (Herceptin)
* epirubicin (Ellence)
* cyclophosphamide (Cytoxan)
* docetaxel (Taxotere)

DETAILED DESCRIPTION:
This is an investigator-initiated, Phase II, non-randomized, single-arm, prospective treatment study. The study will consist of neoadjuvant treatment period (weeks 1 to 20), surgical evaluation period (weeks 20 to 24), and a post-surgical/follow-up period (approximately 3 years). Subjects will be treated on an outpatient basis.

Neoadjuvant therapy will consist of epirubicin + cyclophosphamide given every 2 weeks for four cycles followed by a three week break. Subjects will then receive docetaxel every two weeks for four cycles + trastuzumab (one loading dose) then maintenance dose every 2 weeks for 4 treatments.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant females =/> 18 years of age
* Non-inflammatory breast cancer stage IIA - IIIC or high risk node negative
* Core biopsy of breast demonstrating invasive cancer and documented ER/PgR receptor status
* Normal cardiac function and adequate hematologic function
* Human epidermal growth factor receptor 2 protein (HER2) positive
* No evidence of metastatic disease
* ECOG Performance Status 0 - 1
* Women of childbearing potential must agree to using effective contraception while on treatment and for at least 3 months post-treatment

Exclusion Criteria:

* Treated with other investigational drugs within 30 days
* Uncontrolled intercurrent disease or active infection
* Known sensitivity to e. coli-derived proteins or polysorbate 80
* Psychiatric illness or social situation that would limit study compliance
* Pre-existing peripheral neuropathy > Grade 1
* Cancer within 5 years of screening with the exception of surgically cured nonmelanomatous skin cancer; in-situ carcinoma of the cervix; or in-situ carcinoma of the breast
* Bilateral synchronous breast cancer
* Inflammatory breast cancer
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee S Schwartzberg, MD, FACP, Study Chair — Accelerated Community Oncology Research Network, Inc. (ACORN)
Locations (7):
- United States (7):
  - Advanced Medical Specialties, Miami, Florida
  - Augusta Oncology Associates, Augusta, Georgia
  - Cental Georgia Cancer Care, Macon, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - Hematology Oncology Centers of the Northern Rockies, PC, Billings, Montana
  - Arena Oncology Associates, Great Neck, New York
  - The West Clinic, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 community oncology research sites across the US within the ACORN network participated in this study. Enrollment started in November 2005 and was completed in June 2008.
Pre-assignment Details: Informed consent was obtained from all subjects, and all subjects underwent screening procedures to verify eligibility.
Period: Overall Study
Arm/Group | Neoadjuvant Therapy
Started | 30
Completed | 28
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Therapy
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 50.1 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Able to Complete > 85% of the Planned Dose on Schedule
Description: Feasibility will be determined by evaluating the percentage of subjects able to complete the neoadjuvant portion of the study on time with > 85% of the protocol-specified dose.
Time Frame: From the start of treatment through the neoadjuvant treatment period (approximately 20 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Neoadjuvant Therapy
Number analyzed (Participants) | 30
percentage of participants | 60

2. Primary Outcome: Frequency of Grade 3 or 4 Hematologic and Nonhematologic Toxicities
Description: Toxicities are evaluated according to the Common Terminology Criteria for Adverse Events, version 3.0. Grade refers to the severity of the adverse event (AE). Generally, grade 1 = mild AE; grade 2 = moderate AE; grade 3 = severe AE; grade 4 = life-threatening or disabling AE; grade 5 = death related to AE.
Time Frame: Toxicities are evaluated every 2 weeks during neoadjuvant treatment and assessed once during the post-treatment follow-up period, up to 25 weeks.
Measure: Number; unit: Events
Units Other Than Participants: Events
Arm/Group | Neoadjuvant Therapy
Number analyzed (Participants) | 30
Number analyzed (Events) | 426
Events
  CTCAE grade 3 hematologic events | 2
  CTCAE grade 3 non-hematologic events | 11
  CTCAE grade 4 hematologic events | 0
  CTCAE grade 4 non-hematologic events | 0

3. Secondary Outcome: Pathologic Response
Description: Pathologic response was assessed at time of definitive surgery, scheduled to occur 20-24 weeks after study treatment start. Pathologic complete response was defined as no invasive carcinoma in surgical specimen of breast, but residual ductal carcinoma in situ may be present. Pathologic partial response was defined as >= 50% decrease in sum of diameters in pathologic cancer size compared to pretreatment clinical size. Stable disease was defined as < 50% decrease in sum of diameters in pathologic cancer size compared to pretreatment clinical size, and < 25% increase in sum of diameters.
Time Frame: At completion of neoadjuvant treatment period, up to 24 weeks.
Population: 28 patients went to surgery, so 28 patients were included in the surgery sample. Note that 4 patients in the pathologic complete response (pCR) group had residual ductal carcinoma in situ (DCIS).
Measure: Number; unit: Participants
Arm/Group | Neoadjuvant Therapy
Number analyzed (Participants) | 28
Participants
  Pathologic complete response (pCR) | 16
  Pathologic partial response (pPR) | 9
  Stable disease (SD) | 3

4. Secondary Outcome: Clinical Response Prior to Surgery
Description: Clinical response was assessed via physical exam every 2 weeks during neoadjuvant treatment and via imaging prior to definitive surgery. Clinical complete response was defined as no evidence of cancer in breast by exam or imaging. Clinical partial response was defined as >= 50 % reduction in sum of diameters to measurement of primary lesion compared to pretreatment by exam or imaging. Clinical stable disease was defined as < 50% reduction in sum of diameters to measurement of primary lesion compared to pretreatment by exam or imaging, and < 25% increase in sum of diameters.
Time Frame: Assessed every 2 weeks during neoadjuvant treatment and prior to definitive surgery, up to 23 weeks.
Population: Clinical response assessment was available for 27 patients at the time of surgery.
Measure: Number; unit: Participants
Arm/Group | Neoadjuvant Therapy
Number analyzed (Participants) | 27
Participants
  Clinical complete response | 20
  Clinical partial response | 5
  Clinical stable disease | 2

5. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: LVEF was assessed by echocardiogram (ECHO) or multigated angiogram (MUGA) during neoadjuvant treatment and during follow-up.
Time Frame: At screening, prior to cycle 5, prior to surgery, and then during follow-up at Month 6, 12, 24, and 36
Population: Note that the number of participants analyzed changes with the study interval. At Screening n=30, after Epirubicin/Cyclophosphamide n=30, Pre-surgery n=28, Follow-up Month 6 n=28, Follow-up Month 12 n=20, Follow-up Month 24 n=9, and Follow-up Month 36 n=1.
Measure: Mean (Standard Deviation); unit: LVEF percent
Arm/Group | Neoadjuvant Therapy
Number analyzed (Participants) | 30
LVEF percent
  Screening | 63.55 (7.85)
  After Epirubicin/Cyclophosphamide | 61.94 (6.76)
  Pre-Surgery | 56.88 (10.33)
  Follow-up Month 6 | 57.68 (8.21)
  Follow-up Month 12 | 58.15 (8.47)
  Follow-up Month 24 | 59.38 (3.20)
  Follow-up Month 36 | 55.00 (7.07)

6. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever comes first.
Time Frame: PFS was measured from day 1 of treatment until time of progression or death, whichever comes first, assessed up to 48 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Neoadjuvant Therapy
Number analyzed (Participants) | 29
Months | NA [NA to NA] — Data from 29 patients were included in this analysis, only 3 of whom experienced disease progression. As a result, a median value of PFS could not be estimated. The earliest censored observation occurs at about 15 months.

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from treatment start until death from any cause. The median overall survival time is used to measure OS.
Time Frame: Measured from day 1 of treatment until time of death, assessed up to 48 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Neoadjuvant Therapy
Number analyzed (Participants) | 29
Months | NA [NA to NA] — Data from 29 patients were included in this analysis, only 1 of whom died during the study, an event that occurred about 20 months after start of treatment. As a result, median OS could not be estimated.

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning on day 1 of study treatment until one month after the end of study treatment, up to 25 weeks.
Description: Systematic Assessment - subjects were assessed for adverse events every other week by either the research coordinator, treating physician, or other appropriate sub-investigator.
Arm/Group | Neoadjuvant Therapy
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Therapy (N=30)
Pneumonia (Infections and infestations) | 1
Congestive heart failure (Cardiac disorders) | 1
Medical Error (Injury, poisoning and procedural complications) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Therapy (N=30)
Anemia (Blood and lymphatic system disorders) | 15
Hemoglobin (Blood and lymphatic system disorders) | 1
Myelosuppression (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Congestive heart failure (Cardiac disorders) | 1
Dyspnea (Cardiac disorders) | 3
Ear ache (Ear and labyrinth disorders) | 1
Dry eyes (Eye disorders) | 3
Edema (Eye disorders) | 7
Eye/ear twitching (Eye disorders) | 1
Hyperlacrimation (Eye disorders) | 1
Myelosis (Eye disorders) | 1
Visual changes (Eye disorders) | 1
Watery eyes (Eye disorders) | 11
Abdominal pain.cramps (Gastrointestinal disorders) | 1
Acid reflux (Gastrointestinal disorders) | 4
Difficulty swallowing (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 3
Esophagitis (Gastrointestinal disorders) | 3
Hemorrhage GI Anus (Gastrointestinal disorders) | 1
Gum soreness (Gastrointestinal disorders) | 1
Mouth sores (Gastrointestinal disorders) | 3
Mouth tenderness (Gastrointestinal disorders) | 2
Mucositis (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 22
Stomatitis (Gastrointestinal disorders) | 2
Pain - tooth (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Aches (General disorders) | 2
Chills (General disorders) | 1
Constipation (General disorders) | 6
Cramping bilateral/lower sides (General disorders) | 1
Day sweats (General disorders) | 1
Decreased libido (General disorders) | 1
Diarrhea (General disorders) | 4
Dizziness (General disorders) | 2
Fatigue (General disorders) | 24
Fever (General disorders) | 4
Heartburn (General disorders) | 5
Hot flashes (General disorders) | 6
Malaise (General disorders) | 1
Nose bleed (General disorders) | 2
Pain (General disorders) | 1
Flushing (Immune system disorders) | 1
Herpes simplex (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral thrush (Infections and infestations) | 1
Paranasal sinus reaction (Infections and infestations) | 1
Pulmonary (Infections and infestations) | 1
Sinus infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
ALT (Investigations) | 2
Neutrophils (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Change in appetite (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Weight loss (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Low extremity pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain - back (Musculoskeletal and connective tissue disorders) | 4
Pain - musculoskeletal (Musculoskeletal and connective tissue disorders) | 15
Shoulder/neck soreness (Musculoskeletal and connective tissue disorders) | 1
Weakness (Musculoskeletal and connective tissue disorders) | 4
Neck cyst (Musculoskeletal and connective tissue disorders) | 1
Memory loss (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 6
Pain - headache (Nervous system disorders) | 8
Peripheral paresthesia (Nervous system disorders) | 1
Taste alteration (Nervous system disorders) | 9
Trouble concentrating (Nervous system disorders) | 1
Burning hands and feet (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Daytime insomnia (Psychiatric disorders) | 1
Daytime sleepiness (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 4
Nightmares (Psychiatric disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Irregular menses (Reproductive system and breast disorders) | 1
Menstrual cramps (Reproductive system and breast disorders) | 1
Metromenorrhagia (Reproductive system and breast disorders) | 1
Pain - breast (Reproductive system and breast disorders) | 5
Vaginal dryness (Reproductive system and breast disorders) | 1
Vaginal itching (Reproductive system and breast disorders) | 1
Allergy rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Bilateral crackles (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Sinus problems (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 15
Dry skin (Skin and subcutaneous tissue disorders) | 7
Erythema (Skin and subcutaneous tissue disorders) | 1
Facial rash (Skin and subcutaneous tissue disorders) | 1
Fever blister (Skin and subcutaneous tissue disorders) | 1
Fever blisters (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Itching (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 3
Secondary infection (nails) (Skin and subcutaneous tissue disorders) | 1
Skin pigmentation (Skin and subcutaneous tissue disorders) | 1
Sinus drainage (Surgical and medical procedures) | 1
Hemorrhage pulmonary (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall submit to Aventis for review of confidential information and patent protection purposes, any manuscript or abstract prepared for publication at least 30 days prior to submission to publisher. Upon written request by Aventis to Sponsor within such 30 days, Sponsor agrees to delay such publication until Aventis determines that the publication will not compromise any patent rights. However, such delay shall not exceed 90 additional days.